CLINICAL TRIAL: NCT02465840
Title: The Functional Outcome and Brain Functional MRI of Hand Injury Patients After Different Rehabilitation Programs
Brief Title: Hand Injury Patients Receiving Different Rehabilitation Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CMRPG8D0931
Record Dates: First submitted 2014-12-16; First posted 2015-06-09 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2016-08

CONDITIONS: Hand Injury
Keywords: rehabilitation; functional MRI
MeSH Terms: conditions — Hand Injuries | interventions — Splints; Physical Therapy Modalities; Occupational Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immobilization programs (Placebo Comparator): custom-made protective hand splint physical therapy and occupational therapy
  Interventions: Procedure: custom-made protective hand splint; Other: physical therapy and occupational therapy
- Kleinert programs (Experimental): custom-made dynamic hand splint physical therapy and occupational therapy
  Interventions: Procedure: custom-made dynamic hand splint; Other: physical therapy and occupational therapy

INTERVENTIONS:
Procedure: custom-made dynamic hand splint — custom-made dynamic splinting with more early active exercises intervention.
  Other Names: Dynamic splint
  Arms: Kleinert programs
Procedure: custom-made protective hand splint — Immobilization splint with gentle ROM exercises
  Other Names: resting hand splint
  Arms: Immobilization programs
Other: physical therapy and occupational therapy — both the immobilization and Kleinert programs including physical therapy and occupational therapy for 2-3 times per week.

SUMMARY:
Hand injury is one of common occupational or traumatic injury at outpatient clinic of rehabilitation department. The motor or sensory deficits after hand trauma including bony fracture,tendon / nerve injury, joint stiffness, motion restriction, sensory impairment, or pain lead to impaired upper extremity function, ability for daily activity, or quality of life. Rehabilitation is a kind of therapy for disability after hand trauma. It could provide pain control, improvement of joint motion, stiffness reduction, preventing secondary trauma. The investigators consider that there are some deficits in hand function and range of motion, pain after injury, and some attenuation of brain functional MRI (fMRI) for hand motor control. Therefore, optimal and early intervention of rehabilitation programs may have some benefits for their hand functional outcome and improve the brain activities in fMRI images for the hand motor control.

The aims of this study are to compare the differences in hand motor control area of brain functional MRI (fMRI) between normal subjects and hand injury patients before treatment and to investigate the improvement in brain fMRI activity and functional outcome after early rehabilitation in hand injury patients.

The investigators will collect 40 patients with hand trauma after operation and 10 normal subjects in this study. The 10 normal subjects were allocated in the control group. These 40 patients were randomly divided into 2 experimental groups: 20 patients in group A and 20 patients in group B.

In group A and B, the patients will perform immobilization and Kleinert programs respectively. All patients will perform rehabilitation regimen with 2-3 sessions per week for 3-6 months. Before and after rehabilitation, all patients will receive physical examinations, brain fMRI, and DASH questionnaire for daily activity.

DETAILED DESCRIPTION:
Rehabilitation regimen is a noninvasive therapy for hand injured patients after operation. Protected active/passive motion is the mostly used method. Rehabilitation therapy could provide pain control, improvement of joint motion, stiffness reduction, preventing secondary trauma. The investigators will collect 40 patients with hand trauma after operation and 10 normal subjects in this study. These 40 patients were divided into 2 experimental groups: 20 patients in group A ( immobilization program) and 20 patients in group B (Kleinert program).

A.The immobilization program 0-4 week: dorsal prospective splint in the wrist and MCP joint flexion and IP joint full extension.

3-4 weeks: Hourly: 10 repetitions of passive digital flexion and extension with wrist at 10ﾟextension. Hourly: 10 repetitions of active tendon gliding exercises.

4-6 weeks: dorsal blocking splint discontinued. Gentle blocking exercises initiated 10 repetitions, 4-6 times daily added to passive flexion and tendon gliding.

6-8 weeks: gentle resistive exercise being and progresses gradually. B.The Kleinert program 0-3 day: dorsal protective splint applied with wrist and MCP joints in flexion and IP joints in full extension; elastic traction from fingernail, through palmar pulley, to volar forearm. Velcro strap to allow night release of elastic traction, splinting IPs in full extension.

0-4 weeks: hourly active extension to limits of splint, followed by flexion with elastic traction only. Wound and scar management and education. 4-6 weeks: dorsal protective splint discontinued, sometimes replaced with wrist cuff and elastic traction. Night protective splint to prevent flexion contracture. Active wrist and gentle active fisting initiated unless signs of minimal adhesions. At 6 weeks blocking exercises begin.

6-8 weeks: progressive resistive exercises begin. The investigators will perform the physical examination, brain fMRI, and QuickDASH questionnaire for each patient before the program, 3 and 6 months later. Functional magnetic resonance imaging (fMRI) will be also performed in normal participants.

All patients will perform rehabilitation with 2-3 sessions per week. The investigators will perform the physical examination, brain fMRI, and QuickDASH questionnaire for each patient before the program, 3 and 6 months later. Functional magnetic resonance imaging (fMRI) will be also performed in normal participants.

ELIGIBILITY:
Inclusion Criteria:

* The patients have a hand trauma injury after operation (< 3 months)

Exclusion Criteria:

* previous history of hand injury
* infection disease; arthritis
* systemic neuromuscular disease
* single tendon injury.
* central nerve system disorder

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
change from baseline in motor function | baseline, three months and six months
  QuickDASH quesrtionnaire for upper extremity

SECONDARY OUTCOMES:
Functional MRI | baseline, three months and six months
  "GE" Nuclear Magnetic Resonance Imaging System GE Medical Systems, LLC
wrist pain | baseline, three months and six months
  visual analog scale
wrist sensory | baseline, three months and six months
  light touch, pin prick, position sense
wrist range of motion | baseline, three months and six months
  goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Huang Yu Chi, Bachelor, Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No
no available now

REFERENCES:
- [Background] Vucekovich K, Gallardo G, Fiala K. Rehabilitation after flexor tendon repair, reconstruction, and tenolysis. Hand Clin. 2005 May;21(2):257-65. doi: 10.1016/j.hcl.2004.11.006. PMID 15882604
- [Background] Chesney A, Chauhan A, Kattan A, Farrokhyar F, Thoma A. Systematic review of flexor tendon rehabilitation protocols in zone II of the hand. Plast Reconstr Surg. 2011 Apr;127(4):1583-1592. doi: 10.1097/PRS.0b013e318208d28e. PMID 21187807
- [Background] Karen Pettengill, MS, OTR/L, CHT, Gwendolyn Van Strien, LPT, MSC. Postoperative Management of Flexor Tendon Injuries
- [Background] Diane Cifaldi Collins, Laurie Schwarze, Early progressive resistance following immobilization of flexor tendon repairs. July-September 1991, Pages 111-116
- [Background] Duran RJ, House RG. Controlled passive motion following flexor tendon repairs in zone 2and 3. In: American Academy of Orthopedic Surgeons: Symposium on Tendon Surgery in the Hand. St. Louis : CV Mosby Co.; 1975
- [Background] Iwuagwu FC, McGrouther DA. Early cellular response in tendon injury: the effect of loading. Plast Reconstr Surg. 1998 Nov;102(6):2064-71. doi: 10.1097/00006534-199811000-00038. PMID 9811004
- [Background] Evans RB, Thompson DE. The application of force to the healing tendon. J Hand Ther. 1993 Oct-Dec;6(4):266-84. doi: 10.1016/s0894-1130(12)80328-0. PMID 8124441
- [Background] Bunnell S. Repair of nerves and tendons of the hand. J Bone Joint Surg 1928; 10:1
- [Background] Trumble TE, Vedder NB, Seiler JG 3rd, Hanel DP, Diao E, Pettrone S. Zone-II flexor tendon repair: a randomized prospective trial of active place-and-hold therapy compared with passive motion therapy. J Bone Joint Surg Am. 2010 Jun;92(6):1381-9. doi: 10.2106/JBJS.H.00927. PMID 20516313
- [Background] Tang JB. Clinical outcomes associated with flexor tendon repair. Hand Clin. 2005 May;21(2):199-210. doi: 10.1016/j.hcl.2004.11.005. PMID 15882599
- [Background] Hundozi H, Murtezani A, Hysenaj V, Hysenaj V, Mustafa A. Rehabilitation after surgery repair of flexor tendon injuries of the hand with Kleinert early passive mobilization protocol. Med Arch. 2013;67(2):115-9. doi: 10.5455/medarh.2013.67.115-119. PMID 24341058
- [Background] Tang JB. Indications, methods, postoperative motion and outcome evaluation of primary flexor tendon repairs in Zone 2. J Hand Surg Eur Vol. 2007 Apr;32(2):118-29. doi: 10.1016/J.JHSB.2006.12.009. Epub 2007 Feb 12. PMID 17298858
- [Background] Kleinert HE, Kutz JE, Atasoy E, Stormo A. Primary repair of flexor tendons. Orthop Clin North Am. 1973 Oct;4(4):865-76. No abstract available. PMID 4598164
- [Background] Lister GD, Kleinert HE, Kutz JE, Atasoy E. Primary flexor tendon repair followed by immediate controlled mobilization. J Hand Surg Am. 1977 Nov;2(6):441-51. doi: 10.1016/s0363-5023(77)80025-7. PMID 336675
- [Background] Strickland JW. Flexor tendon injuries. Part 1. Anatomy, physiology, biomechanics, healing, and adhesion formation around a repaired tendon. Orthop Rev. 1986 Oct;15(10):632-45. PMID 3331174
- [Background] Boyer MI, Strickland JW, Engles D, Sachar K, Leversedge FJ. Flexor tendon repair and rehabilitation: state of the art in 2002. Instr Course Lect. 2003;52:137-61. PMID 12690845
- [Background] Angeles JG, Heminger H, Mass DP. Comparative biomechanical performances of 4-strand core suture repairs for zone II flexor tendon lacerations. J Hand Surg Am. 2002 May;27(3):508-17. doi: 10.1053/jhsu.2002.32619. PMID 12015728
- [Background] Xie RG, Zhang S, Tang JB, Chen F. Biomechanical studies of 3 different 6-strand flexor tendon repair techniques. J Hand Surg Am. 2002 Jul;27(4):621-7. doi: 10.1053/jhsu.2002.34311. PMID 12132086
- [Background] Mandeville JB, Rosen BR. Functional MRI. In: Toga AW, MazziottaJC, editors. Brain mapping: the methods. 2nd ed. New York: Academic; 2002. p. 315-49
- [Background] Harel N, Ugurbil K, Uludag K, Yacoub E. Frontiers of brain mapping using MRI. J Magn Reson Imaging. 2006 Jun;23(6):945-57. doi: 10.1002/jmri.20576. PMID 16649202
- [Background] McLarney E, Hoffman H, Wolfe SW. Biomechanical analysis of the cruciate four-strand flexor tendon repair. J Hand Surg Am. 1999 Mar;24(2):295-301. doi: 10.1053/jhsu.1999.0295. PMID 10194013
- [Background] Van der Linden A, Van Camp N, Ramos-Cabrer P, Hoehn M. Current status of functional MRI on small animals: application to physiology, pathophysiology, and cognition. NMR Biomed. 2007 Aug;20(5):522-45. doi: 10.1002/nbm.1131. PMID 17315146
- [Background] Rudin M, Mueggler T, Allegrini PR, Baumann D, Rausch M. Characterization of CNS disorders and evaluation of therapy using structural and functional MRI. Anal Bioanal Chem. 2003 Nov;377(6):973-81. doi: 10.1007/s00216-003-2170-0. Epub 2003 Aug 26. PMID 12942228
- [Background] Tang JB, Wang B, Chen F, Pan CZ, Xie RG. Biomechanical evaluation of flexor tendon repair techniques. Clin Orthop Relat Res. 2001 May;(386):252-9. doi: 10.1097/00003086-200105000-00033. PMID 11347844
- [Background] Sirotakova M, Elliot D. Early active mobilization of primary repairs of the flexor pollicis longus tendon with two Kessler two-strand core sutures and a strengthened circumferential suture. J Hand Surg Br. 2004 Dec;29(6):531-5. doi: 10.1016/j.jhsb.2004.07.002. PMID 15542211
- [Background] Elliot D. Primary flexor tendon repair--operative repair, pulley management and rehabilitation. J Hand Surg Br. 2002 Dec;27(6):507-13. doi: 10.1054/jhsb.2002.0800. No abstract available. PMID 12475505